CLINICAL TRIAL: NCT06294301
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Escalating Single and Multiple Doses of LP-005 in Healthy Volunteers
Brief Title: A Study of Single and Multiple Doses of LP-005 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P10-LP005-01
Record Dates: First submitted 2024-02-03; First posted 2024-03-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Cohort 1: LP-005 Dose 1 (Single) (Experimental)
  Interventions: Biological: LP-005 Dose 1 (Single)
- Cohort 2: LP-005 Dose 2 (Single) (Experimental)
  Interventions: Biological: LP-005 Dose 2 (Single)
- Cohort 3: LP-005 Dose 3 (Single) (Experimental)
  Interventions: Biological: LP-005 Dose 3 (Single)
- Cohort 4: LP-005 Dose 4 (Single) (Experimental)
  Interventions: Biological: LP-005 Dose 4 (Single)
- Cohort 5: LP-005 Dose 5 (Single) (Experimental)
  Interventions: Biological: LP-005 Dose 5 (Single)
- Cohort 6: LP-005 Dose 6 (Single) (Experimental)
  Interventions: Biological: LP-005 Dose 6 (Single)
- Cohort 7: Placebo (Single) (Placebo Comparator)
  Interventions: Biological: Placebo (Single)
- Cohort 8: LP-005 Dose 7 (Multiple) (Experimental)
  Interventions: Biological: LP-005 Dose 7 (Multiple)
- Cohort 9: LP-005 Dose 8 (Multiple) (Experimental)
  Interventions: Biological: LP-005 Dose 8 (Multiple)
- Cohort 10: LP-005 Dose 9 (Multiple) (Experimental)
  Interventions: Biological: LP-005 Dose 9 (Multiple)
- Cohort 11: Placebo (Multiple) (Placebo Comparator)
  Interventions: Biological: Placebo (Multiple)

INTERVENTIONS:
Biological: LP-005 Dose 1 (Single) — A single dose of LP-005 (Dose 1) was administered intravenously.
  Arms: Cohort 1: LP-005 Dose 1 (Single)
Biological: LP-005 Dose 2 (Single) — A single dose of LP-005 (Dose 2) was administered intravenously.
  Arms: Cohort 2: LP-005 Dose 2 (Single)
Biological: LP-005 Dose 3 (Single) — A single dose of LP-005 (Dose 3) was administered intravenously.
  Arms: Cohort 3: LP-005 Dose 3 (Single)
Biological: LP-005 Dose 4 (Single) — A single dose of LP-005 (Dose 4) was administered intravenously.
  Arms: Cohort 4: LP-005 Dose 4 (Single)
Biological: LP-005 Dose 5 (Single) — A single dose of LP-005 (Dose 5) was administered intravenously.
  Arms: Cohort 5: LP-005 Dose 5 (Single)
Biological: LP-005 Dose 6 (Single) — A single dose of LP-005 (Dose 6) was administered intravenously.
  Arms: Cohort 6: LP-005 Dose 6 (Single)
Biological: Placebo (Single) — A single dose of placebo was administered intravenously.
  Arms: Cohort 7: Placebo (Single)
Biological: LP-005 Dose 7 (Multiple) — LP-005 (Dose 7) was administered multiple times intravenously.
  Arms: Cohort 8: LP-005 Dose 7 (Multiple)
Biological: LP-005 Dose 8 (Multiple) — LP-005 (Dose 8) was administered multiple times intravenously.
  Arms: Cohort 9: LP-005 Dose 8 (Multiple)
Biological: LP-005 Dose 9 (Multiple) — LP-005 (Dose 9) was administered multiple times intravenously.
  Arms: Cohort 10: LP-005 Dose 9 (Multiple)
Biological: Placebo (Multiple) — Placebo was administered multiple times intravenously.
  Arms: Cohort 11: Placebo (Multiple)

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, immunogenicity, pharmacokinetics, pharmacodynamics, and efficacy of LP-005 in healthy volunteers. The study will be conducted in 2 parts: Part 1, the single ascending dose (SAD) is the first in human (FIH) study of LP-005 and Part 2, multiple ascending dose (MAD).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged 18 through 50 years
2. Male subjects with a weight of ≥50 kg, female subjects with a weight of ≥45 kg, and BMI between 19.0 and 26.0 kg/m² (inclusive).
3. Vaccination: Meningococcal Conjugate Vaccine, Serogroups A, C, W, Y (MPV-ACYW) meningococcal conjugate vaccine and Streptococcus pneumoniae vaccine should be given 14 days or more before randomisation.
4. Male subjects and their partners or female subjects must agree to use one or more non-pharmaceutical contraceptive methods (such as total abstinence, condoms, Iuds, partner ligation, etc.) during the trial period and for 6 months after the trial, and do not plan to donate sperm or eggs.
5. The subjects fully understand the purpose, nature, method and possible adverse reactions of the experiment, and voluntarily participate in the experiment and sign the informed consent.
6. The subjects were able to communicate well with the researchers and complete the study according to the protocol.

Exclusion Criteria:

1. Participants who are immunocompromised or have one of the following underlying diseases: anatomic absence of spleen (including sickle cell disease); congenital complement component deficiencies (complement component 3 and complement component 4).
2. Any history of Neisseria gonorrhea, meningitis infection, and Guillain-Barré syndrome.
3. Contraindications to meningococcal vaccination (previous medical history such as epilepsy or other brain disorders).
4. Presence or suspicion of active viral, bacterial, fungal, or parasitic infection, including herpes, shingles, or cold sores, within 14 days prior to screening.
5. History of unexplained recurrent infections, or use of systemic antibiotics within 90 days prior to dosing.
6. Malignancy or history of malignancy, except non-melanoma skin cancer cured for more than 3 years.
7. Positive HIV test (HIV-Ab), positive hepatitis B virus (HBV) test (HBsAg), positive hepatitis C virus (HCV), positive anti-syphilis helix-specific antibodies.
8. Participation in a clinical trial of any other drug within 3 months prior to screening or within 5 half-lives of other clinical trial drugs (selecting the longer time period).
9. Women who are pregnant, breastfeeding, or at risk of pregnancy.
10. Any condition deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | Observation for 78 days after administration
  Number of subjects with treatment-related Treatment Emergent Adverse Events (TEAEs).

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) of LP-005 | Observation for 78 days after administration
  The time when the blood drug concentration reaches its peak after a single dose of medication.
Maximum concentration (Cmax) of LP-005 | Observation for 78 days after administration
  The maximum concentration of LP-005 in the bloodstream after administration.
Elimination half-life (t1/2) of LP-005 | Observation for 78 days after administration
  The time required for the concentration of LP-005 in the bloodstream to decrease by half.
Area under the concentration-time curve (AUC0-t) of LP-005 | Observation for 78 days after administration
  The area under the concentration-time curve (AUC) from time zero to the last chosen time point represents the integral of the drug concentration in the bloodstream over the specified duration.
Apparent clearance rate (CL/F) of LP-005 | Observation for 78 days after administration
  The ratio of drug clearance to drug concentration, represents the apparent clearance of a drug after administration, adjusted for bioavailability.
Assessment of immunogenicity | Observation for 78 days after administration
  The proportion of anti drug antibody (ADA) positive subjects at different detection time points.
Assessment of complement C5 activity | Observation for 78 days after administration
  Evaluate complement C5 hemolytic activity and serum concentration of C5 changes from baseline at various time points of assessment.
Assessment of complement C3b activity | Observation for 78 days after administration
  Evaluate C3b deposition on red blood cells and serum concentration of C3b changes from baseline at various time points of assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China